CLINICAL TRIAL: NCT00263094
Title: : An End to the Yom Kippur (and Ramadan) Headache: A Double Blind Placebo Controlled Trial of Prophylactic Rofecoxib in Preventing Ritual Fasting Headache.
Brief Title: An End to the Yom Kippur (and Ramadan) Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SHEBA-04-3395-MD-CTIL
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2006-01-27 (Estimated); Status verified 2006-01

CONDITIONS: Headache
Keywords: Fasting; Headache; Cox 2 Inhibitors; Pain; Prophylaxis
MeSH Terms: conditions — Headache; Fasting; Pain | interventions — rofecoxib

INTERVENTIONS:
Drug: Rofecoxib

SUMMARY:
Fasting is a known trigger for headache. People who fast to comply with religious edict have been shown to be prone to headache which becomes more likely to occur with increasing length of fasting, and in people prone to headache. This has been documented as 'Yom Kippur Headache' and 'First of Ramadan Headache.' We performed a study to test the hypothesis that Rofecoxib, a pain medicine and anti-inflammatory, with a prolonged duration of action would prevent or attenuate headache when taken just prior to the complete (no food or drink) 25 hour fast of Yom Kippur.

DETAILED DESCRIPTION:
Introduction: Religious fasting is associated with headache. This has been documented as 'Yom Kippur Headache' and ' First- of - Ramadan Headache.' The Cox2 inhibitor, rofecoxib, has been reported effective in preventing perimenstrual migraine and in preventing recurrence of migraine. Given its 17 hour half-life, we undertook this study to see whether 50mg rofecoxib taken just prior to the 25 hour Yom Kippur fast would be effective in preventing headache.

Methods: We performed a double blind randomized prospective trial of rofecoxib 50mg vs placebo, taken just prior to the onset of fasting, Yom Kippur 2004. Healthy adults aged 18 - 65 were enrolled from the community and from hospital staff. Subjects completed a demographic data form and questions regarding headache history and a post-fast survey on headache during the fast, headache intensity, general ease of fasting and side effects.

Results: We sent out 170 forms of which 105 were completed and returned. Of those subjects receiving rofecoxib (n=53), ten or 18.9% vs 34 or 65.4 % of the placebo group (n=52) had headache at some point during the fast (p<.0001). Severity of headache in the treatment group was significantly less for the treatment group (3.45 vs 6.29 on a visual analog scale of 10 (p = .009)). None of those receiving rofecoxib reported a 'more difficult than usual fast' whereas the distribution of difficult to easy fast among the placebo group was more even.

Conclusion: Rofecoxib 50mg taken prior to a twenty five hour ritual fast prevents and attenuates fasting headache.

ELIGIBILITY:
Inclusion Criteria:

* History of fasting headache
* Age 18-65
* Intention to fast on Yom Kippur
* History of Fasting on Yom Kippur

Exclusion Criteria:

* Pregnant or Nursing Women
* Known allergy to NSAID type medication
* History of chronic illness including heart, kidney, liver or peptic ulcer disease, hypertension, diabetes, lung disease including asthma, or a history of gastrointestinal bleeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-09; Study Completion 2004-11

PRIMARY OUTCOMES:
Reduction in incidence of headache during fast in treatment group versus control group

SECONDARY OUTCOMES:
Reduction in severity of headache in treatment versus control groups.
General ease of fast in treatment vs control groups

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Drescher, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Mosek A, Korczyn AD. Yom Kippur headache. Neurology. 1995 Nov;45(11):1953-5. doi: 10.1212/wnl.45.11.1953. PMID 7501139
- [Background] Awada A, al Jumah M. The first-of-Ramadan headache. Headache. 1999 Jul-Aug;39(7):490-3. doi: 10.1046/j.1526-4610.1999.3907490.x. PMID 11279933
- [Background] Von Seggern RL, Mannix LK, Adelman JU. Rofecoxib in the prevention of perimenstrual migraine: an open-label pilot trial. Headache. 2004 Feb;44(2):160-5. doi: 10.1111/j.1526-4610.2004.04033.x. PMID 14756855